CLINICAL TRIAL: NCT06145828
Title: Clinical Application of Cytokine Adsorption Technology in AIDS Patients With Severe Pneumonia and/or Septic Shock: An Observational Study.
Brief Title: Clinical Application of Cytokine Adsorption Technique in AIDS Patients With Severe Pneumonia and/or Septic Shock
Status: Recruiting | Type: Observational
Sponsor: Guangzhou 8th People's Hospital (Other)
Responsible Party: Principal Investigator, Linghua LI, Chief physician, Guangzhou 8th People's Hospital
Other Study IDs: 202322259
Record Dates: First submitted 2023-11-14; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: AIDS Pneumonia; Septic Shock
Keywords: AIDS; Severe Pneumonia; Septic Shock; Cytokine Adsorption Technique
MeSH Terms: conditions — Shock, Septic; Acquired Immunodeficiency Syndrome; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cytokine Adsorption Combined with Standard Treatment Group: This group receives cytokine adsorption combined with standard treatment, specifically via hemoperfusion using the standard 211 protocol: two hemoperfusions within the first 24 hours, followed by one hemoperfusion daily. Each hemoperfusions session does not exceed 6 hours, lasting a total of 3 days. All patients also undergo blood perfusion treatment with the addition of a plasma separator.
  Interventions: Device: Cytokine Adsorption
- Standard Treatment Group: This group receives only standard treatment . Standard treatment includes symptomatic supportive therapy, etiological therapy, fluid resuscitation, application of vasopressors, and non-invasive or invasive ventilation therapy.

INTERVENTIONS:
Device: Cytokine Adsorption — During treatment with cytokine adsorption cartridge, the patient's blood is passed through these cartridges, which contain substances that can adsorb specific cytokines. Excess cytokines are captured and removed by these substances, and then the cleansed blood is returned to the patient's body.
  Groups: Cytokine Adsorption Combined with Standard Treatment Group

SUMMARY:
Observing the Real-World Application Effectiveness of Cytokine Immune Adsorption Technology in AIDS Patients with Severe Pneumonia or septic shock.

DETAILED DESCRIPTION:
This is a prospective, single-center, non-randomized, clinical observational cohort study primarily focused on observing the clinical effects of cytokine adsorption technology in patients with AIDS complicated by severe pneumonia and/or septic shock. Based on the real-world application of cytokine adsorption technology in AIDS patients with severe pneumonia or septic shock, the study divides patients into two groups: one receiving cytokine adsorption combined with standard treatment, and another receiving standard treatment only. The study aims to observe the impact of these two different treatment strategies on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV infection;
2. Progression to AIDS stage: CD4+ count <200 cells/ul and/or occurrence of AIDS opportunistic infections;
3. Age between 18 and 65 years;
4. Meeting the diagnosis of severe pneumonia or septic shock:

   1. The criteria for severe pneumonia diagnosis refer to the 2021 ATS (American Thoracic Society) and IDSA (Infectious Diseases Society of America) guidelines for the treatment of community-acquired pneumonia;
   2. The criteria for septic shock refer to the Chinese Society of Critical Care Medicine's "Chinese Guidelines for the Emergency Treatment of Sepsis/Septic Shock (2018).

Exclusion Criteria:

1. Coexisting central nervous system lesions, severe liver disease, or cirrhosis;
2. Concurrent AIDS-related or unrelated tumors;
3. Women who are pregnant or breastfeeding;
4. Severe underlying diseases of the heart, lungs, liver, kidneys, etc.;
5. Alcohol abuse or drug use;
6. The researcher believes that the overall condition of the subject affects the evaluation and completion of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study participants come from the OSPWH (Patients With HIV/AIDS) cohort at the Guangzhou Eighth People's Hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-10-23 (Estimated); Study Completion 2027-10-23 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 4 weeks
  Compare the mortality rates of the cytokine adsorption combined with standard treatment group and the standard treatment group.

SECONDARY OUTCOMES:
Improvement in critical care scoring | Baseline and during treatment at weeks 1, 2, 3, 4.
  Improvements in the intensive care scoring systems SOFA score and APACHE II score from baseline and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Linghua Li, PhD, Study Chair — Guangzhou Eighth People's Hospital
Locations (1):
- Guangzhou Eighth People's Hospital, Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Pei F, Yao RQ, Ren C, Bahrami S, Billiar TR, Chaudry IH, Chen DC, Chen XL, Cui N, Fang XM, Kang Y, Li WQ, Li WX, Liang HP, Lin HY, Liu KX, Lu B, Lu ZQ, Maegele M, Peng TQ, Shang Y, Su L, Sun BW, Wang CS, Wang J, Wang JH, Wang P, Xie JF, Xie LX, Zhang LN, Zingarelli B, Guan XD, Wu JF, Yao YM; Shock and Sepsis Society of Chinese Research Hospital Association; China Critical Care Immunotherapy Research Group; International Federation of the Shock Societies (IFSS). Expert consensus on the monitoring and treatment of sepsis-induced immunosuppression. Mil Med Res. 2022 Dec 26;9(1):74. doi: 10.1186/s40779-022-00430-y. PMID 36567402
- [Result] Wendel Garcia PD, Hilty MP, Held U, Kleinert EM, Maggiorini M. Cytokine adsorption in severe, refractory septic shock. Intensive Care Med. 2021 Nov;47(11):1334-1336. doi: 10.1007/s00134-021-06512-0. Epub 2021 Sep 1. No abstract available. PMID 34471938